CLINICAL TRIAL: NCT03626259
Title: Effect of the Administration of Losartan / Amlodipine in Fixed Combination Versus Losartan on Hemodynamic and Arterial Stiffness Parameters in Patients With Systemic Hypertension Grade 1 and 2
Brief Title: Losartan/Amlodipine on Hemodynamics Parameters and Arterial Stiffness in Arterial Hypertension
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centro Universitario de Ciencias de la Salud, Mexico (Other)
Responsible Party: Principal Investigator, Fernando Grover Paez, Principal Investigator, Centro Universitario de Ciencias de la Salud, Mexico
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CUCS-INTEC-MV-LOAM-001
Record Dates: First submitted 2018-08-08; First posted 2018-08-10 (Actual); Last update posted 2018-08-17 (Actual); Status verified 2018-08

CONDITIONS: Hypertension
Keywords: hypertension; losartan/amlodipine; arterial stiffness
MeSH Terms: conditions — Hypertension | interventions — amlodipine-losartan drug combination; Losartan

STUDY DESIGN:
Intervention Model Description: assignment
Who Masked: Participant, Investigator
Masking Description: double blind (subject, investigator)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- losartan and amlodipine (Other): Individuals with SAH grade 1 or 2 without triple pharmacological therapy.
  Interventions: Drug: Losartan and Amlodipine
- Losartan (Active Comparator): Individuals with SAH grade 1 or 2 without triple pharmacological therapy.
  Interventions: Drug: Losartan

INTERVENTIONS:
Drug: Losartan and Amlodipine — Losartan and amlodipine in fixed combination capsules, 100mg/5mg. One time daily with the first bite of eat meal per 8 weeks
  Other Names: Bicartial
  Arms: losartan and amlodipine
Drug: Losartan — Losartan capsules, 100mg. One time daily with the first bite of eat meal per 8 weeks
  Arms: Losartan

SUMMARY:
Systemic Arterial Hypertension (SAH) is a disease with a high prevalence in Mexico and worldwide. SAH is associated with an increase in cardiovascular morbidity and mortality, causing cardiovascular disease (CVD), heart failure (HF), as well as chronic kidney disease (CKD). Several of the physiopathological mechanisms observed are: the increase in cardiac output, central aortic pressure (CAP), pulse wave velocity (PWV) and peripheral vascular resistance (PVR), which leads to the generation of damage to the target organ. The identification not only of the peripheral arterial pressure, but also of these hemodynamic parameters and arterial stiffness would allow a better cardiovascular characterization of the patients. However, the measurements of hemodynamic parameters and arterial stiffness can vary during the 24 hours from individual to individual by all known mechanisms involved in the regulation of blood pressure such as cortisol, central nervous system, the peripheral nervous system, along with the renin angiotensin and aldosterone system, which are usually only measured in a single moment. Generally, the choice of drug in a patient with SAH is based only on the values of peripheral blood pressure at the time of the measurement. The use of oscillometric equipment such as the Mobil-O-Graph 24 allows to the investigators to know the hemodynamic and arterial stiffness behavior during 24 hours; therefore, this could favor the choice of the most appropriate antihypertensive drug, dose and administration time. The use of angiotensin II receptor antagonists (ARA II) At1 blockers such as losartan and calcium channel blockers (CCB) for instance amlodipine have shown a reduction in CAP and peripheral blood pressure respectively in patients with SAH. The most prescribed drugs in health units worldwide are enalapril, amlodipine, losartan and atenolol, of which the most used combination is losartan with amlodipine. There are no studies to date that allow investigators to identify the effect of the administration of losartan / amlodipine in a fixed combination form on the hemodynamic parameters and arterial stiffness of patients with SAH. Therefore, the objective of the present study is to evaluate the effect of this fixed combination versus losartan on hemodynamic and arterial stiffness parameters based on the behavior of these for 24 hours.

DETAILED DESCRIPTION:
In the present investigation the investigators expect to know the effect of the administration of losartan / amlodipine in fixed combination versus losartan on hemodynamic parameters and arterial stiffness in patients with arterial hypertension grade 1 and 2. For this purpose the investigators will conduct a double-blind randomized trial, each group will be compose by 14 male and female patients, 40-65 years old, with hypertension, neither with diabetes nor being under triple pharmacological therapy. Randomization will determine who will receive the intervention during an 8- week trial (losartan/amlodipine in fixed combination capsule, 100mg/5mg 1 time daily or losartan capsule 100mg 1 time daily). The clinical findings and laboratory tests include a metabolic profile and biosafety, which will be at baseline and by the 8th week . Body weight, body fat, body mass index (BMI) and blood pressure will be determined during the initial and final visit, in addition to hemodynamics parameters of arterial stiffness like cardiac output, central aortic pressure (CAP), pulse wave velocity (PWV) and peripheral vascular resistance (PVR) by an oscillometric monitoring system via Mobil-O -Graph® 24. Adverse events and adherence to treatment will be documented. Statistical analysis: Mann-Whitney U Test and Wilcoxon exact test. It is considered with significance at p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of hypertension grade 1 or 2 according to the criteria of the American Heart Association (2017)
* Written informed consent
* Patients who are undergoing antihypertensive treatment and who, at the trial of the investigator and taking care of the health and safety of the patient, can undergo at least 2 weeks of washing prior to the visit of day 0 (it will be evaluated on a case-by-case basis).

Exclusion Criteria:

* Systolic blood pressure ≥ 180 mmHg or diastolic blood pressure ≥120 mmHg
* Diabetes Mellitus
* Treated with triple pharmacological therapy
* Untreated thyroid disease
* Total cholesterol >400mg/dl
* Triglycerides >400mg/dl
* Liver enzymes (alt and ast) more tan twice the normal range
* Glomerular filtration rate <60ml/min (Cockcroft-Gault)

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2018-08-06 (Actual); Primary Completion 2019-01-15 (Estimated); Study Completion 2019-06-14 (Estimated)

PRIMARY OUTCOMES:
Pulse Wave Velocity (PWVao) | 56 days
  Before and after intervention with oscillometric monitoring system via Mobil-O -Graph® 24. Maximum score 12 m/s

SECONDARY OUTCOMES:
Peripheral vascular resistance | 56 days
  Before and after intervention with oscillometric monitoring system via via Mobil-O -Graph®. Maximum score 1.8s*mmHg/ml
Cardiac output | 56 days
  Before and after intervention with oscillometric monitoring system via via Mobil-O -Graph®. Maximum score 6.5L/min
Pulse Pressure (PP) | 56 days
  Before and after intervention with oscillometric monitoring system via via Mobil-O -Graph® 24. Maximun score <75 mmHg
Augmentation Index (AIx) | 56 days
  Before and after intervention with oscillometric monitoring system via via Mobil-O -Graph® 24. Maximum score 110%
Systolic blood pressure | 56 days
  Before and after intervention using a digital manometer. Maximum score 160 mmHg
Diastolic blood pressure | 56 days
  Before and after intervention using a digital manometer. Maximum score 100 mmHg
Creatinine | 56 days
  Before and after intervention by spectrophotometry. Maximum score 1.3 mg/dl

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Grover Paez, PhD, Principal Investigator — Institute of Experimental and Clinical Therapeutics (INTEC), CUCS, University of Guadalajara
Locations (1):
- Institute of Experimental and Clinical Therapeutics (INTEC), CUCS, University of Guadalajara, Guadalajara, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: No